CLINICAL TRIAL: NCT04974450
Title: Effect of Trigona Honey to Intestinal Microbiota, Lipid Profile and Anthropometric Status in Obese Individuals
Brief Title: Trigona Honey and Intestinal Microbiota Among Obese People
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hasanuddin University (Other)
Responsible Party: Principal Investigator, Bumi Herman, Assistant Lecturer, Hasanuddin University
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1007210708
Record Dates: First submitted 2021-07-14; First posted 2021-07-23 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Obesity
Keywords: obesity; trigona honey; lipid profile; microbiota; anthropometry
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Two different groups will be given two different honey. In the intervention group, trigona honey will be administered for 8 weeks whereas the control group will be given artificial honey that has a similar taste and appearance to the intervention group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Masking in terms of taste and appearance is applied to yield a similar product. Researchers prepare artificial honey formula with citrus flavor to mimic the natural taste of trigona honey. Neither the care provider nor the investigator aware of the allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trigona Honey (Experimental): The intervention will be given by oral route in a form of liquid of 70-gram trigona honey once daily for 8 weeks
  Interventions: Dietary Supplement: Trigona honey
- Control (Active Comparator): The intervention will be given by oral route in a form of liquid of 70-gram artificial honey once daily for 8 weeks
  Interventions: Dietary Supplement: control

INTERVENTIONS:
Dietary Supplement: Trigona honey — composition : vitamin C 0.15%, Protein 1.32%, lipid 0.23%, carbohydrate 64.12%, beta carotene 10.61 ppm, Calcium 273,23, magnesium 338.94, zinc 12.49 ppm, and acidity 5.76. Total polyphenol 133.52 ppm, total flavonoid 159.62 ppm. This liquid has a sour profile
  Arms: Trigona Honey
Dietary Supplement: control — Artificial honey with fructose, Glucose, pure honey (2,271%), citric acid, and lime extract (0,076%).
  Arms: Control

SUMMARY:
Objective :

Nutrition intervention is one of the approaches to deal with obesity. Natural honey with its polyphenol component has an impact on the intestinal microbiota and lipid profile. Intestinal microbiota such as lactobacillus and bifidobacteria produce exopolysaccharide which plays important roles against obesity. This research aims to assess the effect of Trigona biroi honey on body mass index, lipid profile, and microbiota profile

Design A Quasi-experimental study involving two arms (trigona honey) and control will be conducted. The outcome of interests are body mass index, lipid profile, and microbiota profile

Hypothesis using superiority trial, trigona honey will

1. improve microbiota (increase lactobacillus and bifidobacteria and reduce clostridium)
2. Improving lipid profile
3. lowering body mass index

DETAILED DESCRIPTION:
Target population :

This study will recruit healthy participants with a body mass index of more than 27

allocation : non-random with propensity score matching

Arms

1. Trigona honey (intervention) composition : vitamin C 0.15%, Protein 1.32%, lipid 0.23%, carbohydrate 64.12%, beta carotene 10.61 ppm, Calcium 273,23, magnesium 338.94, zinc 12.49 ppm, and acidity 5.76. Total polyphenol 133.52 ppm, total flavonoid 159.62 ppm. This liquid has a sour profile
2. Active comparator Commercial honey with fructose, Glucose, pure honey (2,271%), citric acid, and lime extract (0,076%).

Intervention 8 weeks, once daily. This also applied to the control group

Outcome :

1. Microbiota detected using Polymerase Chain Reaction (PCR)

   1. Sample: Stool
   2. extraction with 70% ethanol primary PCR
   3. primer (Lactobacillus and bifidobacteria)
2. Lipid Profile using blood plasma and homogenous assay High-Density Lipoprotein, Low-Density Lipoprotein, Triglyceride, total cholesterol
3. Anthropometry Body mass index, body composition (fat percentage), waist circumference

Sample Size was calculated using the difference of HDL between groups with the following parameters :

Effect size =0.3 Type 1 error = 5% Power of Study = 80% dropout = 20% total participant 336

Analysis Intention to treat will be applied. The descriptive statistic will be used to describe the baseline characteristic of participants. The bivariate analysis will be conducted to see the association of demographic factors to the outcome. If the matching of the participant yields a similar baseline characteristic, the difference of mean between the two groups will be analyzed using an independent t-test. Otherwise, linear mixed model will be applied

ELIGIBILITY:
Inclusion Criteria:

1. Defined as obese with a body mass index of more than 27
2. Not having a gastrointestinal disease
3. Not allergic to the honey component

Exclusion criteria:

1. Consuming probiotics for a minimum of one month
2. Consuming antibiotics for a minimum of one month

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Level of intestinal microbiota in stool | Changes of microbiota level from day 0 to day 60 after intervention
  the level of bifidobacteria, clostridium, and lactobacillus (in colony factor unit/grams) in stool measured using polymerase chain reaction

SECONDARY OUTCOMES:
Body Mass Index | Changes of body mass index from day 0 to day 60 after intervention
  measured by dividing body weight in kilogram per square meter of height
Lipid Profile | Changes of lipid profile from day 0 to day 60 after intervention
  the level of High-Density Lipoprotein, Low-density lipoprotein, total cholesterol and triglyceride in blood plasma

CONTACTS AND LOCATIONS:
Overall Officials: Andi S Rahma, MD, Principal Investigator — Hasanuddin University
Locations (1):
- Wahidin Sudirohusodo General Hospital, Makassar, South Sulawesi, Indonesia

IPD SHARING:
Plan to Share IPD: No
de-identified data will be shared accordingly

REFERENCES:
- [Background] de Melo FHC, Menezes FNDD, de Sousa JMB, Dos Santos Lima M, da Silva Campelo Borges G, de Souza EL, Magnani M. Prebiotic activity of monofloral honeys produced by stingless bees in the semi-arid region of Brazilian Northeastern toward Lactobacillus acidophilus LA-05 and Bifidobacterium lactis BB-12. Food Res Int. 2020 Feb;128:108809. doi: 10.1016/j.foodres.2019.108809. Epub 2019 Nov 21. PMID 31955768
- [Background] Jiang L, Xie M, Chen G, Qiao J, Zhang H, Zeng X. Phenolics and Carbohydrates in Buckwheat Honey Regulate the Human Intestinal Microbiota. Evid Based Complement Alternat Med. 2020 Feb 26;2020:6432942. doi: 10.1155/2020/6432942. eCollection 2020. PMID 32184894
- [Background] Lashani E, Davoodabadi A, Soltan Dallal MM. Some probiotic properties of Lactobacillus species isolated from honey and their antimicrobial activity against foodborne pathogens. Vet Res Forum. 2020 Spring;11(2):121-126. doi: 10.30466/vrf.2018.90418.2188. Epub 2020 Jun 15. PMID 32782740
- [Background] Mohd Rafie AZ, Syahir A, Wan Ahmad WAN, Mustafa MZ, Mariatulqabtiah AR. Supplementation of Stingless Bee Honey from Heterotrigona itama Improves Antiobesity Parameters in High-Fat Diet Induced Obese Rat Model. Evid Based Complement Alternat Med. 2018 Nov 21;2018:6371582. doi: 10.1155/2018/6371582. eCollection 2018. PMID 30643535
- [Background] Samat S, Kanyan Enchang F, Nor Hussein F, Wan Ismail WI. Four-Week Consumption of Malaysian Honey Reduces Excess Weight Gain and Improves Obesity-Related Parameters in High Fat Diet Induced Obese Rats. Evid Based Complement Alternat Med. 2017;2017:1342150. doi: 10.1155/2017/1342150. Epub 2017 Jan 26. PMID 28246535